CLINICAL TRIAL: NCT02009865
Title: A 12-Week, Randomized, Double-Blind, Olive Oil-Controlled Phase 3 Study to Assess the Efficacy and Safety of EPANOVA™ in Subjects With Severe Hypertriglyceridemia (EVOLVE II)
Brief Title: Epanova® for Lowering Very High Triglycerides II (EVOLVE II)
Acronym: EVOLVEII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5880C00001; OM-EPA-011 (Other: AstraZeneca Plc)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia; Dyslipidemia; Eicosapentaenoic acid; EPA; Docosahexaenoic acid; DHA
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epanova 2 g/day (Experimental): Arm 1
  Interventions: Drug: Epanova
- Olive Oil 2 g/day (Placebo Comparator): Arm 2
  Interventions: Drug: Olive Oil

INTERVENTIONS:
Drug: Epanova — Epanova will be provided in 1 g polyacrylate-coated soft gel capsules. Two capsules will be taken once per day, without regard to meals, for 12 weeks. At clinic visits, study drug will be administered at the clinic after fasting blood draws are complete.
  Other Names: omega-3 free fatty acids
  Arms: Epanova 2 g/day
Drug: Olive Oil — Olive oil will be provided in 1 g polyacrylate-coated soft gel capsules. Two capsules will be taken once per day, without regard to meals, for 12 weeks. At clinic visits, study drug will be administered at the clinic after fasting blood draws are complete.
  Other Names: placebo comparator
  Arms: Olive Oil 2 g/day

SUMMARY:
This is a double-blind, randomized, olive oil-controlled study to investigate the efficacy and safety of Epanova as an adjunct therapy to diet for reduction of TG levels in subjects with severe hypertriglyceridemia. The study consists of an approximately 8-week screening period that includes a diet and lifestyle stabilization and washout period and a 12-week treatment period.

DETAILED DESCRIPTION:
[During the screening period and treatment period, all visits are to be within ±3 days of the scheduled time.]

Screening Period:

Visit 1 will occur at Week -8 for subjects requiring washout and/or statin, cholesterol-absorption inhibitor (CAI), or statin-CAI stabilization. This includes subjects who:

* Were previously on omega-3 drugs/supplements;
* Require adjustment to or addition of permitted statins, CAI, or statin-CAI combination;
* Have not been on a permitted stable dose of statin, CAI, or statin-CAI combination for at least 4 weeks prior to Visit 1; and/or
* Need to washout of bile acid sequestrants, fibrates, niacin, and other supplements known to alter lipid metabolism.

For these subjects who require washout and/or statin, CAI, or statin-CAI stabilization, at Visit 1 (Week -8) screening procedures will be performed. Subjects will return at Visit 1a (Week -2) for their first qualifying lipid measurement.

For subjects not requiring washout, Visit 1 will occur at Week -2. All screening procedures will be performed at this visit including the first qualifying lipid measurement.

At Visit 2 (Week -1), all subjects will return for their second lipid qualifying measurement. If at Visit 2 the subject does not have an average TG ≥500 mg/dL (6 mmol/L) and <2500 mg/dL (28 mmol/L), the TG measurement may be repeated one additional time after Visit 2 (Visit 2a). The subject's qualifying measurement would be the average of Visit 1 or 1a + Visit 2 + Visit 2a (repeat measurement).

To be eligible for randomization, the subject must have a qualifying TG ≥500 mg/dL (6 mmol/L) and <2500 mg/dL (28 mmol/L). Of the total number of subjects, approximately 50% will have a qualifying TG >885 mg/dL (10 mmol/L) and <2500 mg/dL (28 mmol/L). Once approximately 50% of the total subjects has been reached for each TG group, enrollment of subjects with that specific TG criterion will stop. Subjects will be equally allocated to each treatment group.

[At the screening visit, all subjects will receive counseling regarding the National Cholesterol Education Program (NCEP) Therapeutic Lifestyle Changes (TLC) diet and will receive basic instructions on how to follow this diet. See Appendix C.]

Treatment Period:

At Visit 3 (Week 0), approximately 116 subjects will be randomized in a 1:1 ratio to receive daily olive oil 2 g or Epanova 2 g. Subjects will be stratified by lipid-altering drugs to ensure a balanced allocation of subjects who are users and non-users of the following permitted lipid-altering drugs in each treatment group: statin, CAI, or statin-CAI combination. During the treatment period, subjects will return to the site at Visit 4 (Week 6), Visit 5 (Week 10), and Visit 6 (Week 12) for efficacy and safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding of the study procedures, willingness to adhere to the study schedule, and agreement to participate in the study by giving written informed consent prior to screening;
2. Willing to use an appropriate and effective method of contraception;
3. Qualifying (average of Visit 1 or 1a + Visit 2 + Visit 2a [repeat measurement]) serum TG ≥500 mg/dL (6 mMol/L) and <2500 mg/dL (28 mMol/L);
4. Body mass index ≥20 kg/m2;
5. Untreated dyslipidemia or dyslipidemia treated with a statin, CAI, or statin-CAI combination that has been stable for 6 weeks prior to randomization; and
6. Willingness to maintain current physical activity level and follow the TLC diet throughout the study.

Exclusion Criteria:

1. Allergy or intolerance to omega-3 fatty acids, omega-3-acid ethyl esters, or fish;
2. Known lipoprotein lipase impairment;
3. Known non-responder to omega-3 or fenofibrate therapy;
4. Use of any prescription medications containing EPA and/or DHA (eg, Lovaza® or Vascepa®) within 8 weeks prior to randomization. Up to 1 g capsule/day of an omega-3 dietary supplement will be permitted;
5. Unable to discontinue use of bile acid sequestrants, fibrates or niacin (other than niacin-containing vitamins <200 mg), or any supplement used to alter lipid metabolism including but not limited to dietary fiber supplements, red rice yeast supplements, garlic supplements, soy isoflavone supplements, sterol/stanol products, or policosanols at screening;
6. Use of tamoxifen, estrogens, or progestins that has not been stable for >4 weeks at screening or is unstable prior to randomization;
7. Use of oral or injected corticosteroids or anabolic steroids prior to randomization;
8. History of hospitalization for pancreatitis in the last 5 years;
9. Uncontrolled diabetes (hemoglobin A1c [HbA1c] >10%);
10. Uncontrolled hypothyroidism or thyroid-stimulating hormone (TSH) >5 mIU/L;
11. History of cancer (other than basal cell carcinoma) in the past 2 years;
12. Cardiovascular event (ie, myocardial infarction, acute coronary syndrome, new onset angina, stroke, transient heart attack, unstable congestive heart failure requiring a change in treatment), revascularization procedure or vascular surgery within 6 months of randomization;
13. Use of simvastatin 80 mg or Vytorin 10/80 mg;
14. Recent history (within 6 months of randomization) of significant nephrotic syndrome, pulmonary, hepatic, biliary, gastrointestinal, or immunologic disease;
15. Poorly controlled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
16. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × the upper limit of normal (ULN); if ALT/AST is >3 × ULN, the levels have been stable for 3 months and are <5 × ULN;
17. Exposure to any investigational product within 4 weeks of randomization; or
18. Any condition or therapy which, in the opinion of the Investigator, might pose a risk to the subject or make participation in the study not in the subject's best interest.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2014-12-23 (Actual); Study Completion 2014-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (14):
  - Research Site, Los Angeles, California
  - Research Site, St. Petersburg, Florida
  - Research Site, Addison, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
- Research Site, Chicoutimi, Quebec, Canada
- Czechia (3):
  - Research Site, Hradec Kralova
  - Research Site, Trutnov
  - Research Site, Zlín
- Denmark (4):
  - Research Site, Esbjerg
  - Research Site, Gentofte Municipality
  - Research Site, Herlev
  - Research Site, Viborg
- Hungary (7):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Sátoraljaújhely
  - Research Site, Székesfehérvár
  - Research Site, Szikszó
- Netherlands (2):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was planned at 43 sites, and in total, 162 were randomized in a 1:1 ratio to two treatment groups, Epanova (n=81) and Olive Oil (n=81). Randomization of subjects was stratified by two factors: 1. use of lipid-altering drugs (yes, no), and 2. Qualifying triglycerides values below or above 885 mg/dL.
Pre-assignment Details: In total, 379 subjects were screened from the 43 sites.
Groups:
- Epanova; Olive Oil: 2g once daily (QD)
Period: Overall Study
Arm/Group | Epanova | Olive Oil
Started | 81 | 81
Completed | 80 | 76
Not Completed | 1 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epanova | Olive Oil | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (10.60) | 50.0 (10.88) | 50.2 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 65 | 62 | 127
Lipid-altering drug use [Number; unit: Participants]
  Yes | 36 | 37 | 73
  No | 45 | 44 | 89
At least 1 qualifying TG category > 885 mg/dL [Number; unit: Participants]
  Yes | 53 | 52 | 105
  No | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Triglyceride for All Subjects
Description: This primary endpoint was tested in parallel together with the first of the secondary endpoints, each at 0.025 Type I error rate.
Time Frame: From Baseline to Week 12 Endpoint
Population: Full Analysis Set (FAS)
Measure: Median (Inter-Quartile Range); unit: Percentage of change (%)
Arm/Group | Epanova | Olive Oil
Number analyzed (Participants) | 81 | 81
Percentage of change (%) | -28.1 [-42.1 to -5.5] | -10.2 [-36.4 to 23.0]
Statistical Analysis 1: Comparison: Epanova vs Olive Oil; Missing values were imputed using probabilities of missing estimated from logistic regression; Test type: Superiority or Other; p = 0.017, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -14.2, 95% CI 2-sided [-26.2 to -2.8] — The estimated median difference and its 95% CI were based on Hodges Lehmann procedure

2. Secondary Outcome: Percent Change in Triglycerides for Subjects With at Least 1 Qualifying Triglyceride >885 mg/dL
Description: This first secondary endpoint in subjects with at least 1 qualifying triglyceride >885 mg/dL was tested in parallel together with the primary endpoint, each at 0.025 Type I error rate.
Time Frame: From Baseline to Week 12 Endpoint
Population: FAS
Measure: Median (Inter-Quartile Range); unit: Percentage of change (%)
Arm/Group | Epanova | Olive Oil
Number analyzed (Participants) | 53 | 52
Percentage of change (%) | -37.5 [-46.1 to -18.1] | -9.3 [-36.3 to 27]
Statistical Analysis 1: Comparison: Epanova vs Olive Oil; Main analysis with missing values imputed using probabilities of missing estimated from logistic regression; Test type: Superiority or Other; p = 0.0008, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -26.3, 95% CI 2-sided [-40.5 to -11.5] — The estimated median difference and its 95% CI were based on Hodges Lehmann procedure

3. Secondary Outcome: Percent Change in Non-High-Density Lipoprotein Cholesterol (mg/dL)
Description: This secondary endpoint, together with the 3rd. and 4th secondary ones, was treated as the core secondary, and the p value from the hypothesis test on its treatment comparison was adjusted by using Hommel's procedure.
Time Frame: From Baseline to Week 12 Endpoint
Population: FAS
Measure: Median (Inter-Quartile Range); unit: Percentage of change (%)
Arm/Group | Epanova | Olive Oil
Number analyzed (Participants) | 81 | 81
Percentage of change (%) | -8.8 [-15.7 to -1.4] | 0.4 [-13.5 to 14.2]
Statistical Analysis 1: Comparison: Epanova vs Olive Oil; Missing values were imputed using probabilities of missing estimated from logistic regression; Test type: Superiority or Other; p = 0.0180, Wilcoxon (Mann-Whitney) — Adjusted by using Hommel's procedure; Median Difference (Final Values) = -9.0, 95% CI 2-sided [-14.8 to -2.8] — The estimated median difference and its 95% CI were based on Hodges Lehmann procedure

4. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol (mg/dL)
Description: This secondary endpoint, together with the 2nd. and 4th. secondary ones, was treated as the core secondary, and the p value from the hypothesis test on its treatment comparison was adjusted by using Hommel's procedure.
Time Frame: From Baseline to Week 12 Endpoint
Population: FAS
Measure: Median (Inter-Quartile Range); unit: Percentage of change (%)
Arm/Group | Epanova | Olive Oil
Number analyzed (Participants) | 81 | 81
Percentage of change (%) | 3.4 [-5.1 to 12.5] | 3.1 [-6.3 to 10.9]
Statistical Analysis 1: Comparison: Epanova vs Olive Oil; Missing values were imputed using probabilities of missing estimated from logistic regression; Test type: Superiority or Other; p = 0.7117, Wilcoxon (Mann-Whitney) — Adjusted by using Hommel's procedure; Median Difference (Final Values) = -0.3, 95% CI 2-sided [-3.5 to 4.9] — The estimated median difference and its 95% CI were based on Hodges Lehmann procedure

5. Secondary Outcome: Percent Change in Triglyceride(mg/dL) in Subjects With Biochemically Defined Fredrickson Type V (Triglyceride/Very-Low-Density Lipoprotein Cholesterol ≥6)
Description: This secondary endpoint in subjects with Biochemically Defined Fredrickson Type V (Triglyceride/Very-Low-Density Lipoprotein Cholesterol ≥6), together with the 2nd. and 3rd.secondary ones, was treated as the core secondary, and the p value from the hypothesis test on its treatment comparison was adjusted by using Hommel's procedure.
Time Frame: From Baseline to Week 12 Endpoint
Population: FAS
Measure: Median (Inter-Quartile Range); unit: Percentage of change (%)
Arm/Group | Epanova | Olive Oil
Number analyzed (Participants) | 55 | 57
Percentage of change (%) | -24.7 [-43.3 to -2.8] | -12.4 [-38.8 to 14.2]
Statistical Analysis 1: Comparison: Epanova vs Olive Oil; Missing values were imputed using probabilities of missing estimated from logistic regression; Test type: Superiority or Other; p = 0.3034, Wilcoxon (Mann-Whitney) — Adjusted by using Hommel's procedure; Median Difference (Final Values) = -10.3, 95% CI 2-sided [-23.9 to 3.5] — The estimated median difference and its 95% CI were based on Hodges Lehmann procedure

ADVERSE EVENTS:
Arm/Group | Epanova | Olive Oil
Serious Adverse Events (participants affected / at risk) | 1/81 | 2/81
Other Adverse Events (participants affected / at risk) | 29/81 | 28/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova (N=81) | Olive Oil (N=81)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova (N=81) | Olive Oil (N=81)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (6)
Eructation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
All (Gastrointestinal disorders) | 12 (17) | 7 (15)
ALL (Infections and infestations) | 10 (11) | 6 (7)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (2) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
ALL (Nervous system disorders) | 5 (5) | 3 (6)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
ALL (Investigations) | 4 (5) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Gastric pH decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2)
ALL (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
ALL (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinitis allergi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALL (General disorders) | 3 (3) | 2 (3)
Fatigue (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
ALL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
ALL (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ALL (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
ALL (Cardiac disorders) | 1 (1) | 1 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
ALL (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
ALL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ALL (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ALL (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
ALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No